CLINICAL TRIAL: NCT06137326
Title: Efficacy of Pulsed Electromagnetic Field Therapy Versus Laser Acupuncture on Female Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: PEMF vs Laser for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Director of Electromyography lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEMF-LAS-2023
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized controlled trial with two arms receiving different interventions.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Electromagnetic Field Therapy (Experimental)
  Interventions: Device: Pulsed Electromagnetic Field Therapy
- Laser Acupuncture (Active Comparator)
  Interventions: Device: Laser Acupuncture

INTERVENTIONS:
Device: Pulsed Electromagnetic Field Therapy — Participants in this arm will receive pulsed electromagnetic field (PEMF) therapy to the pelvic floor area along with pelvic floor muscle training. The PEMF device generates a pulsed magnetic field with the following parameters: frequency 10 Hz, intensity 200 μT, pulse duration 250 μs. It will be applied over the pelvic floor for 20 minutes per session, 5 days per week for 8 weeks.
  Arms: Pulsed Electromagnetic Field Therapy
Device: Laser Acupuncture — Participants in this arm will receive low-level laser acupuncture to pelvic floor trigger points along with pelvic floor muscle training. A continuous wave 810 nm diode laser will be used at 100 mW power and 0.5 J/point, delivered to 6 pelvic floor acupoints bilaterally (12 points total) for 15 seconds per point. Acupuncture will be performed 3 days per week for 8 weeks.
  Arms: Laser Acupuncture

SUMMARY:
Stress urinary incontinence, or involuntary urine leakage during activities like coughing, laughing, or exercise, is a common condition that impacts quality of life for many women. Pelvic floor muscle training is often used to treat stress incontinence, but additional therapies may enhance outcomes. This randomized controlled trial will compare two physical therapy modalities, pulsed electromagnetic field (PEMF) therapy versus laser acupuncture, along with pelvic floor training for improving stress urinary incontinence in 60 adult women. The study will evaluate their effects on pelvic floor muscle strength, severity of urine leakage, and quality of life. We hypothesize that PEMF and laser acupuncture will both improve stress incontinence, but PEMF will be more effective based on greater pelvic floor stimulation. The study aims to provide evidence on these physical therapy options so that optimized treatment plans can be developed for women with stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 18-65 years with stress urinary incontinence
* Able to comply with study procedures and schedule

Exclusion Criteria:

* Prior pelvic floor surgery
* Pregnancy
* Active urinary tract infection
* Pelvic organ prolapse >Stage 2
* Neurologic disorder affecting urinary function

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Change in pelvic floor muscle strength | Baseline and 8 weeks
  elvic floor muscle strength will be assessed using a calibrated perineometer device that measures vaginal squeeze pressure. Strength will be recorded in cm H2O.

SECONDARY OUTCOMES:
Change in Severity Index for urinary incontinence | Baseline and 8 weeks
  Severity of urine leakage will be scored using the Severity Index (SI), a validated index that rates leakage frequency and volume on a 0-20 point scale. Higher scores indicate greater severity.
Change in ICIQ-UI SF score | Baseline and 8 weeks
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a validated quality of life questionnaire for urinary incontinence. It contains 3 scored items, with total score range of 0-21. Higher scores denote greater impact on QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamada, Ph.D, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided